CLINICAL TRIAL: NCT07273682
Title: A Nurse-facilitated Interdisciplinary Transitional Care Programme for Childhood Cancer Survivors and Their Parents to Improve Symptom Management: a Feasibility Randomised Waitlist-controlled Trial
Brief Title: Nurse-led Transitional Care to Improve Symptom Management in Childhood Cancer Survivors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Eva Ho, associate professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: nurse-facilitated care
Record Dates: First submitted 2025-11-19; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-10

CONDITIONS: Pediatric Cancer
Keywords: Omaha system; nurse-facilitated; interdisciplinary transitional care programme; Chinese childhood cancer survivors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Other: Counseling based on Omaha system
- Wait-list control group (Other)
  Interventions: Other: Counseling based on Omaha system; Other: Usual Care

INTERVENTIONS:
Other: Counseling based on Omaha system — Investigators developed the intervention based on the Omaha system and investigators' previous studies. The intervention will last for 12 weeks. During week 1, dyads (a pairing of a child with their parent) will have a 1-hour face-to-face consultation with a RN. The RN will assess every dyad using the Omaha system to identify any problems. The Omaha system covers 42 problems grouped into 4 categories, including environmental, physiological, psychosocial and health-related behaviours. After identifying the problems, the RN will deliver corresponding interventions according to the intervention scheme in the Omaha system. Subsequent follow-up will be provided by the RN via zoom during weeks 2, 3, 4, 6, 8, 10 and 12 to evaluate their progress in terms of knowledge, behaviour and status using the rating scale in the Omaha system. The RN will assign further interventions, based on the Omaha system, to address their specific needs. Each follow-up should last around 30 minutes.
Other: Usual Care — Dyads in this group will receive usual care, defined as the existing care practices provided by the hospital, which include a discharge checklist and educational materials regarding the care. After the completion of data collection for all timepoints, they will be invited to join the counselling based on Omaha system intervention.
  Arms: Wait-list control group

SUMMARY:
This study aims to evaluate the feasibility and preliminary effectiveness of a nurse-facilitated interdisciplinary transitional care programme, based on the Omaha system, for Chinese childhood cancer survivors (CCSs) and their parents in Hong Kong. Investigators will conduct a two-arm, randomized waitlist-controlled trial at the Hong Kong Children's Hospital, the only local center for CCS follow-up. Sixty-eight dyads (CCS aged 13-18 and a parent) will be randomized to either the 12-week nurse-led intervention or usual care. The intervention includes an initial face-to-face assessment and regular follow-ups via Zoom, focusing on symptom management, health education, and self-care empowerment, with referrals to other professionals as needed. The control group receives standard discharge care and educational materials, and will be offered the intervention after data collection. Outcomes will be assessed at baseline, and 3 and 6 months post-intervention, including symptom management, quality of life, caregiver burden, self-efficacy, and emergency department visits. Feasibility will be evaluated by recruitment, retention, attendance, and data completeness rates. If effective, this programme could improve transitional care and symptom management for CCSs and their families, and inform clinical practice and policy in Hong Kong and beyond.

ELIGIBILITY:
Inclusion Criteria for CCSs:

* aged between 13 and 18 years
* diagnosed with any cancer
* completion of active cancer treatment within a month
* communicate in Chinese

Inclusion Criteria for parents:

* mother or father who has a significant caregiving role in the child's life
* could participate in the intervention at the same time as their child
* communicate in Chinese
* have an electronic device to access zoom

Exclusion Criteria for CCSs:

* cognitive impairment
* social and/or behavioural problem
* have terminal cancer
* participate in any similar intervention

Exclusion Criteria for parents:

* severe emotional problems
* participate in any similar intervention

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Screening rate | Baseline
  Number of dyads screened divided by number of dyads available for screening.
Eligibility rate | Baseline
  Number of dyads eligible divided by number of dyads screened.
Recruitment rate | Baseline
  Number of eligible dyads agree to join divided by number of eligible dyads.
Randomization rate | Baseline
  Number of dyads being randomized divided by number of participating dyads.
Intervention attendance rate | Immediately after the intervention completion
  Number of dyads who complete the intervention divided by number of dyads in the intervention group.
Retention rate | Baseline, immediately after the intervention completion, 3 months after intervention completion, 6 months after intervention completion
  Number of dyads remaining in the study divided by number of dyads being randomized.
Completion rate | Baseline, immediately after the intervention completion, 3 months after the intervention completion, 6 months after the intervention completion
  Number of dyads who complete the questionnaire divided by number of questionnaires distributed.
Missing data | Baseline, immediately after the intervention completion, 3 months after the intervention completion, 6 months after the intervention completion
  Percentage of missing data
Adverse events | During the study period including 12-week intervention and 6 months follow-up
  Number of unfavourable events and/or worsening reported.

SECONDARY OUTCOMES:
Cancer-related symptoms in CCSs | Baseline, immediately after the intervention completion, 3 months after the intervention completion, 6 months after the intervention completion
  It will be used to assess the cancer-related symptoms in CCSs. It has 30 items in seven domains: nutrition-related, psychosocial/central nervous system, oropharyngeal, bone marrow toxicity/neuropathy, skin/other toxicities, neurotoxicity and respiratory/other. Each item will be evaluated on a five-point scale, from 0 to 4. The psychometric properties have been well validated in CCSs.
CCSs' quality of life (QoL) | Baseline, immediately after the intervention completion, 3 months after the intervention completion, 6 months after the intervention completion
  Paediatric Quality of Life Questionnaire (PedsQoL) will be used to assess the CCSs' QoL. It comprises 23 items. CCSs will rate their experience during the preceding month on a five-point scale. All items will be reverse-scored and linearly transformed onto a 0-100-point scale. This scale has well-established psychometric properties in CCSs.
Caregiver burden of parents | Baseline, immediately after the intervention completion, 3 months after the intervention completion, 6 months after the intervention completion
  The caregiver burden in parents will be assessed using the Chinese version of the Caregiver burden inventory (CBI), which consists of 24 items in five dimensions: time-dependence, development, physical, social and emotional burdens. Each item will be evaluated from 0 (not at all relevant) to 4 (very relevant), with the total score between 0 and 96. The Chinese version is a valid and reliable instrument for use.
Caregiving competence of parents | Baseline, immediately after the intervention completion, 3 months after the intervention completion, 6 months after the intervention completion
  Caregiving competence scale (CCS) will be used to record the competence of parents regarding their caregiving. This scale comprises four items, each of which is evaluated on a four-point rating scale, from 1 (not at all) to 4 (very much). The psychometric properties of the Chinese version have been well established.
Parental quality of life (QoL) | Baseline, immediately after the intervention completion, 3 months after the intervention completion, 6 months after the intervention completion
  Parental QoL will be assessed using the Chinese version of the EQ-5D, with one question regarding each of five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The values will be weighted to convert into a value from 1 (full health) to 0 (equivalent to being dead). The psychometric properties of the EQ-5D have been well validated in the Chinese population.
Number of emergency department (ED) visits | During the study period including 12-week intervention and 6 months follow up
  It will be assessed by number of walk-in visits to the emergency department. These data will be collected in the central medical system with the assistance of PI in HKCH (Hong Kong Children's Hospital).